CLINICAL TRIAL: NCT01071642
Title: The Influence of Angiotensin Converting Enzyme Inhibitors and Angiotensin Receptor Blockers on Renal Function in Patients Undergoing Non-emergent Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Talya Wolak, senior doctor internal medicine department, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sor495209ctil
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Blood Pressure
Keywords: Change in eGFR from baseline to 72 hours following the exposure to the contrast.; Rate of eGFR decrease>25% from the baseline; Length of hospitalization.; Requirement of unplanned therapy for elevated blood pressure

ARMS (3):
- continue ace-i and arb's versus dicontinue (No Intervention)
- group b (Active Comparator)
  Interventions: Drug: stop ace-i/arb 24 h before procedure and restarted 24 hours after the procedure
- group c (Active Comparator)
  Interventions: Drug: ACE/ARB stopped 24 hours before procedure and start immediately after

INTERVENTIONS:
Drug: stop ace-i/arb 24 h before procedure and restarted 24 hours after the procedure — ACE/ARB stopped 24 hours prior to the procedure and restarted 24 hours after the procedure
  Arms: group b
Drug: ACE/ARB stopped 24 hours before procedure and start immediately after — ACE/ARB stopped 24 hours prior to the procedure and restarted immediately after the procedure
  Arms: group c

SUMMARY:
The aim of the current study is to evaluate prospectively whether concomitant administration of RAAS blockers (namely ACE-I and ARBs') influence the change in estimated GFR (eGFR) after administration of contrast media in patients undergoing non-emergent coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age>18 years
* 2. Subjects on chronic therapy with ACE-I and/or ARBs' (confirmed by electronic records in their medical file)
* 3. Subjects planned to undergo non-emergent coronary angiography.
* 4. Signed informed consent

Exclusion Criteria:

* 1. eGFR<30 ml/min at baseline
* 2. Chronic utilization of NSAIDS and Cox-2 selective inhibitors
* 3. Chronic treatment with mineralocorticosteroid receptor blocker
* 4. Systolic blood pressure<90 mmHg
* 5. Planned staged (repeated) procedure within 48 hours
* 6. Administration of contrast within 14 days prior to the enrollment
* 7. contraindication to stop ACE-I or ARB'S

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in eGFR from baseline to 48 hours following the exposure to the contrast. | 48 hours after exposure to the contrast

SECONDARY OUTCOMES:
1. Rate of eGFR decrease>25% from the baseline, 2. Length of hospitalization, | 48-72 hours after exposure to contrast

CONTACTS AND LOCATIONS:
Locations (1):
- Talya Wolak, Bear Sheva, Israel